CLINICAL TRIAL: NCT05554484
Title: A Multi-center, Controlled, Open, Phase I Clinical Trial to Assess the Safety of AMI-DC (Autologous Dendritic Cells) Treatment in Patients With Acute Anterior Wall ST-segment Elevation Myocardial Infarction Who Received Reperfusion by Primary Percutaneous Coronary Intervention (PCI)
Brief Title: AMI-DC in Patients With Anterior Wall Myocardial Infarction
Acronym: AMI-DC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Kiyuk Chang, MD,PhD, Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMI-DC
Record Dates: First submitted 2022-09-02; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Stage A (Sequential allocation): 6 for experimental group, 3 for control group Stage B (Randomized allocation): 9 for experimental group, 12 for control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AMI-DC (Experimental): Infusion of AMI-DC + Guideline directed optimal medical therapy
  Interventions: Biological: Autologous peripheral blood-derived tolerogenic dendritic cells
- Standard treatment (No Intervention): Control, Guideline directed optimal medical therapy

INTERVENTIONS:
Biological: Autologous peripheral blood-derived tolerogenic dendritic cells — AMI-DC, autologous dendritic cell product Inject 7.5 x 106 cells hypodermically to 1~4 sites in the left axillary lymph node between 5-7 days after PCI and 12-14 days after PCI. . The administration must be done within 30 minutes after fully liquified.
  Arms: AMI-DC

SUMMARY:
The purpose of this trial is to assess the safety of AMI-DC treatment. The participants who voluntarily sign the consent form will be screened according to the inclusion/exclusion criteria then allocated either to the experimental group (drug therapy and AMI-DC therapy) or to the control group (drug therapy only). Both the experimental group and the control group are treated with standard medical therapy after PCI. The experimental group will be hospitalized for 4-5 days after 1st injection, and 1 day after 2nd injection. Vital signs are collected after 30 minutes, 1 hour, 2 hours and 4 hours after the 1st and 2nd injections and the subjects will be monitored 24 hours for safety assessment. The identical examination will also be performed in the control group and the results will be collected.

DETAILED DESCRIPTION:
The registration of study subjects follows two stages (stages A & B). In Stage A, 6 subjects in the experimental group and 3 subjects in the control group will sequentially be registered, then will be monitored for 10 weeks to assess safety. If Stage A passes the safety assessment, the rest will be recruited and randomly allocated to either experimental or control group in Stage B.

Approximately 300cc of whole blood will be collected only from patients assigned to the experimental group. The amount of blood collection can be supervised and adjusted at the discretion of the investigators. Collected blood will be cultured for 4 days to generate the dendritic cells. Then, 5~10x106 cells are administered subcutaneously at 1-4 sites in the left axillary regions between 5-7 days after PCI and between 12-14 days after PCI.

Echocardiography and cardiac MRI will be examined for any signs of adverse reaction to ensure safety and evaluate cardiac functions at baseline and after 6 months.

* In stage A, 6 people are sequentially allocated to the experimental group and 3 people are sequentially allocated to the control group.
* The experimental group are monitored for 10 weeks following the 2nd AMI-DC to assess safety. Stage B is implemented once determined safe to proceed.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers who qualify all the following conditions

  1. Between the ages 19 through 80

     Patients within 24 hours from primary PCI with a diagnosis of acute anterior wall ST-segment elevation myocardial infarction and systolic dysfunction:

     acute myocardial infarction patient with an electrocardiogram (12-lead ECG) result corresponding to any of the following (ST-segment elevation 0.1 mV in two or more limb leads or 0.2 mV elevation in two or more contiguous precordial leads)
  2. Left ventricular ejection fraction (LVEF) below 50% by echocardiography
  3. Hemodynamically stable (SBP >100 mmHg, HR <110 bpm, SO2 >95%)
  4. Able-bodied for collection of approximately 300cc of blood for generation of autologous dendritic cells who qualify the following conditions
* Body weight: 50 kg or above for men, 45 kg or above for women
* Hb level of 12.0 g/dL or above 5) Signed the written consent form for this clinical trial

Exclusion Criteria:

* Volunteers who correspond to any of the following conditions

  1. LV thrombus
  2. Difficulty in accessing femoral artery for sheath insertion due to peripheral artery disease
  3. Previous history of PCI, CABG due to myocardial infarction
  4. Renal failure: serum Creatinine >2.5 mg/dL
  5. Acute or chronic infections
  6. Known contraindications to MRI
  7. Hemorrhagic disorders (PT INR >2)
  8. History of malignant tumor within 5 years
  9. A life expectancy of 1 year or less
  10. Tested positive with HIV, HBV, HCV and/or syphilis
  11. Autoimmune disease
  12. Pregnant or nursing mothers
  13. Participated in other clinical trials within past 30 days
  14. Deemed unfit for this clinical trial by the investigators
  15. Disagreed to use an approved method of contraception (Men: vasectomy, double diaphragm, or effective contraception used by the partner. Women: IUD, IUS or hormonal contraceptives) during the trial period.
  16. Moderate-to-severe liver disease (ALT is more than 5 times the upper limit of normal)
  17. Acute myocardial infarction patients at high bleeding risk with Hb 11g/dL or more Use or are scheduled to use oral anticoagulants for a long period of time Spontaneous hemorrhage that required hospitalization or blood transfusion within the past 6 months Thrombocytopenia (platelet count of <100x109/L) Liver cirrhosis with portal hypertension Severe ischemic stroke within the past 6 months, with spontaneous intracerebral hemorrhage and cerebrovascular malformation Major surgery or severe injury within the past 30 days

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-07 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Outcome 1 | Up to 6 months
  Occurrence of Ventricular Arrhythmias, Perforation, Myocardial Ischemia, or Any sign of infection that occur during the entire study period
Primary Safety Outcome 2 | Week 12
  Occurrence of Ventricular Arrhythmia or Bradyarrhythmia in 24-hour Holter monitoring at 12 weeks.
Primary Efficacy Outcome | up to 6 months
  Cumulated incidence ratio of MACE (death from any cause, HF admission, VT/VF, stroke) at 6 months

SECONDARY OUTCOMES:
Change in infarct size | up to 6 months
  Change in infarct size measured by MRI between the baseline and 6 months.
Change in left ventricular ejection fraction | up to 6 months
  Changes in left ventricular ejection fraction (in percent) by echocardiography/MRI between the baseline and 6 months.
Change in LV chamber | up to 6 months
  Changes in left ventricular end-systolic (milliliter)/end-diastolic volume (milliliter) measured by echocardiography/MRI between the baseline and 6 months.
Change in LV wall motion | up to 6 months
  Changes in WMSI measured by echocardiography/MRI between the baseline and 6 months.
Change in polarization of lymphocyte by FACS | up to 12 weeks
  Changes in polarization of lymphocyte by FACS (in percentage) at baseline (before the 1st AMI-DC administration), before the 2nd AMI-DC administration, at 3 weeks, and at 12 weeks.
Change in serum cytokine | up to 12 weeks
  Changes in IL-1, TNF-a, IL-6, and IL-10 (in picogram per milliliter) by ELISA at baseline (before the 1st AMI-DC administration), before the 2nd AMI-DC administration, at 3 weeks, and at 12 weeks.
Change in white blood cell count | up to 6 months
  Changes in white blood cell count, neurtrophil count, and lymphocyte (number per liter) count between the baseline and 6 months.
Change in C-reactive protein (CRP) | up to 6 months
  Changes in CRP (milligram per liter) between the baseline and 6 months.
Change in NT-proBNP | up to 6 months
  Changes in NT-pro-BNP (picogram per liter) between the baseline and 6 months.
Change in patients' HF symptom | up to 6 months
  Changes in NYHA functional class at each visit

CONTACTS AND LOCATIONS:
Locations (1):
- Eun Ho Choo, Seoul, South Korea